CLINICAL TRIAL: NCT02273908
Title: Patient-reported-outcomes(PROs) in Chronic Low Back Pain Patients With Accompanying Lower Limb Pain (Neuropathic Component) Treated With Pregabalin in Primary Care Settings
Brief Title: PROs in Chronic Low Back Pain Patients With Accompanying Lower Limb Pain (Neuropathic Component) Treated With Pregabalin
Acronym: PRO
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0081333
Record Dates: First submitted 2014-10-17; First posted 2014-10-24 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2016-10

CONDITIONS: Low-Back Pain
Keywords: Low-Back Pain; Neuropathic Pain; Pregabalin
MeSH Terms: conditions — Low Back Pain; Neuralgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pregabalin: Patients will be treated for 8 weeks with pregabalin in primary care: no intervention
  Interventions: Other: No intervention
- Usual care: Patients will be treated for 8 weeks with other analgesics in usual care: no intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — The study is observational

SUMMARY:
The purpose of this study is to evaluate the effect of pregabalin comparing with the conventional analgesic care in chronic low back pain patients with accompanying lower limb pain (neuropathic component) treated in primary care settings under routine clinical practice.

DETAILED DESCRIPTION:
Rational and background :

The care for low back pain associated with neuropathic pain is a problem often encountered in daily outpatient.

And the care effectiveness has been frequently evaluated by the patients directly, because the pain would be felt by patients themselves.

On the view of those, we decided to investigate the clinical treatment outcome of pregabalin or other analgesics medication for relief of pain and improvement of sleep interference and QOLs by Patient-reported outcomes.

Research question and objectives :

To evaluate the effect of pregabalin comparing with the conventional analgesic care in chronic low back pain patients with accompanying lower limb pain (neuropathic component) treated in primary care settings under routine clinical practice.

Study design:

This is an 8-week, multicenter prospective observational study. Subjects who have chronic low back pain patients with accompanying lower limb pain (with a neuropathic component) and meet all other entry criteria are enrolled at baseline in the duration of study. The analgesic treatment is determined by the clinical judgment of the physician in charge of patient management. This therapeutic choice is not related to the decision to take part in the study. All enrolled subjects will be received with analgesic treatment. The study requires 3 visits at least, baseline/enrollment visit, Week 4 visit and Week 8 visit (or discontinuation).

ELIGIBILITY:
Inclusion Criteria:

1. Subject who received the enough study information and signed informed consent form.
2. Subject who had chronic low back pain accompanying with lower limb pain from the knee to the ankle.
3. Subject is male or female patient ≥18 years old.
4. Subject who has complained low back pain for 3 months or more before Visit 1.
5. Subject who is refractory to prior analgesics for 3 months and more.
6. Subject who is able and willing to complete all study related assessment and comply with the study schedule and clinical procedures at clinic.
7. Subject whose pain Numeric Rating Scale(NRS) ≥ 5 at baseline (based on recall over the past week)

Exclusion Criteria:

1. Subject who, in the opinion of the investigator, was not likely to complete the trial for whatever reason.
2. Subject who has been already treated by pregabalin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic low-back pain patients with neuropathic component will be treated with pregabalin or other analgesics
Sampling Method: Non-Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Fujii, MD, Study Director — Director of Pain/Neuroscience Medical Affairs,Pfizer Japan Inc.
Locations (33):
- Japan (33):
  - Kimura Clinic, Nagoya, Aichi-ken
  - Jin Orthopaedic Clinic, Ichikawa, Chiba
  - Satoh Orthopaedic Clinic, Ichikawa, Chiba
  - Shiraishi Orthopaedic Clinic, Ichikawa, Chiba
  - Ota General Hospital, Kawasaki, Kanagawa
  - Aoki Orthpaedic Clinic, Sagamihara, Kanagawa
  - Hiyoshi Hocho Clinic, Yokohama, Kanagawa
  - Yamamoto Memorial Hospital, Yokohama, Kanagawa
  - Ageo Medical Clinic, Ageo, Saitama
  - Arai Orthopaedic Clinic, Fujimino, Saitama
  - Nakaicho Clinic, Adachi City, Tokyo
  - Mitsuda Orthopaedic Clinic, Chiyoda City, Tokyo
  - Kyobashi Orthopaedic Clinic, Chūō, Tokyo
  - Morishima Clinic, Edogawa City, Tokyo
  - Kita Akabane Orthopaedic Clinic, Kita-ku, Tokyo
  - Takeuchi Orthopaedic Clinic, Kita-ku, Tokyo
  - Tanaka Orthopaedic Clinic, Koganei, Tokyo
  - Araki Clinic, Koto, Tokyo
  - Kohsei Chuo General Hospital, Meguro City, Tokyo
  - Meguro Seikeigeka Naika, Meguro City, Tokyo
  - Meguro Yuai Clinic, Meguro City, Tokyo
  - Takemoto Orthopaedic Clinic, Ohta, Tokyo
  - Shiotani Pain Clinic, Shinagawa, Tokyo
  - Daido Hospital, Toshima City, Tokyo
  - Senkawa Shinoda Orthopaedic Clinic, Toshima City, Tokyo
  - Takahashi Orthopaedic Clinic, Toshima City, Tokyo
  - Kanazawa Hospital, Kanazawa, Yokohama
  - Katayama Orthopaedic Memorial Hospital, Tsurumi, Yokohama
  - Nakamura Orthopaedic Clinic, Kagoshima
  - Showa-kai Clinic, Kagoshima
  - Clinic Ushitani, Miyazaki
  - Kohnan Matsumoto Orthopaedic Clinic, Miyazaki
  - Iwasaki Orthopaedic Clinic, Saitama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Taguchi T, Igarashi A, Watt S, Parsons B, Sadosky A, Nozawa K, Hayakawa K, Yoshiyama T, Ebata N, Fujii K. Effectiveness of pregabalin for the treatment of chronic low back pain with accompanying lower limb pain (neuropathic component): a non-interventional study in Japan. J Pain Res. 2015 Aug 5;8:487-97. doi: 10.2147/JPR.S88642. eCollection 2015. PMID 26346468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was conducted from Jun. 2014 to Dec. 2014 at 33 study sites.
Groups:
- Pregabalin: Patients will be treated for 8 weeks with pregabalin in primary care:no intervention
- Other Analgesics: Patients will be treated for 8 weeks with other analgesics in usual care:no intervention
Period: Overall Study
Arm/Group | Pregabalin | Other Analgesics
Started | 157 | 174
Completed | 124 | 169
Not Completed | 33 | 5
Not completed — Adverse Event | 16 | 0
Not completed — Lost to Follow-up | 10 | 1
Not completed — Did not meet entrance criteria | 3 | 2
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Pregabalin: Patients will be treated for 8 weeks with pregabalin in primary care :no intervention
- Other Analgesics: Patients will be treated for 8 weeks with other analgesics in usual care :no intervention
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Other Analgesics | Total
Number analyzed (Participants) | 157 | 174 | 331
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 44 | 87
  >=65 years | 114 | 130 | 244
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (14.12) | 70.7 (12.17) | 70.0 (13.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 106 | 198
  Male | 65 | 68 | 133
Region of Enrollment [Number; unit: participants]
  Japan | 157 | 174 | 331

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain Related Sleep Interference Scale (PRSIS - Past Week Recall)
Description: The Pain Related Sleep Interference Scale (past week recall) consists of an 11-point rating scale ranging from 0 (pain did not interfere with sleep) to 10 (pain completely interfered with sleep). Change the rating scale from baseline to week 8 in each group. Subjects are to describe how their pain has interfered with their sleep during the past week by choosing the appropriate number between 0 and 10.
Time Frame: Baseline, Final Visit (Week 8)
Population: Full Analysis Set; consisted of subjects who had at least one evaluable observation from any of the patient-reported outcomes, and only evaluable subjects who contributed to the particular outcome were evaluated in each analysis. 'n' signifies number of participants who were evaluable for specified categories at different time points
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin | Other Analgesics
Number analyzed (Participants) | 137 | 172
scores on a scale
  Baseline (n=137,172) | 3.1 (2.63) | 2.9 (2.40)
  Change from baseline at Week 8 (n=115,160) | -1.306 (0.197) | -0.357 (0.168)
Statistical Analysis 1: Comparison: Pregabalin vs Other Analgesics; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -0.949, 95% CI 2-sided [-1.459 to -0.439]

2. Secondary Outcome: Change From Baseline in Roland Morris Disability Questionnaire (RMDQ)-Total Score-
Description: The RMDQ is an index of how well patients with low back pain are able to function with regard to daily activities. The score for the index ranges from 0 to 24 with a lower score indicating better function.
Time Frame: Baseline, Visit2 (Week4), Final Visit (Week8 or discontinuation)
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin | Other Analgesics
Number analyzed (Participants) | 137 | 172
scores on a scale
  Baseline (n=137,172) | 10.8 (5.20) | 9.1 (4.90)
  Change from baseline at Week 4(n=118,160) | -2.893 (0.312) | -1.006 (0.270)
  Change from baseline at Week 8 (n=115,160) | -3.670 (0.335) | -1.411 (0.287)
Statistical Analysis 1: Comparison: Pregabalin vs Other Analgesics; Analysis on the mean difference between two groups with the change from baseline at Week 8; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -2.259, 95% CI 2-sided [-3.131 to -1.387]
Statistical Analysis 2: Comparison: Pregabalin vs Other Analgesics; Analysis on the mean difference between two groups with the change from baseline at Week 4; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.887, 95% CI 2-sided [-2.704 to -1.071]

3. Secondary Outcome: Change From Baseline in Roland Morris Disability Questionnaire (RMDQ)-Japanese Standardized Score-
Description: as for outcome 2
Time Frame: Baseline, Visit2 (Week4), Final Visit (Week8 or discontinuation)
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin | Other Analgesics
Number analyzed (Participants) | 113 | 138
scores on a scale
  Baseline (n=113,138) | 39.77 (12.453) | 44.92 (9.845)
  Change from baseline at Week 4 (n=97,128) | 5.1062 (0.6905) | 2.3772 (0.6039)
  Change from baseline at Week 8 (n=99,127) | 6.8377 (0.6833) | 3.5359 (0.6040)
Statistical Analysis 1: Comparison: Pregabalin vs Other Analgesics; Analysis on the mean difference between two groups with the change from baseline at Week 8; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 3.3018, 95% CI 2-sided [1.4903 to 5.1133]
Statistical Analysis 2: Comparison: Pregabalin vs Other Analgesics; Analysis on the mean difference between two groups with the change from baseline at Week 4; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Least square mean difference = 2.7290, 95% CI 2-sided [0.9047 to 4.5533]

4. Secondary Outcome: Change From Baseline in Pain Numeric Rating Scale (Pain NRS - Past Week Recall)
Description: The Pain NRS (past week recall) consists of an 11-point numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst possible pain). Subjects are asked to describe their average pain during the past week by choosing the appropriate number between 0 and 10.
Time Frame: Baseline, Visit2 (Week4), Final Visit (Week8 or discontinuation)
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin | Other Analgesics
Number analyzed (Participants) | 137 | 172
scores on a scale
  Baseline (n=137,172) | 6.2 (1.17) | 5.8 (1.14)
  Change from baseline at Week 4 (n=118,160) | 1.763 (0.172) | -1.089 (0.149)
  Change from baseline at Week 8 (n=115,160) | -2.166 (0.181) | -1.336 (0.155)
Statistical Analysis 1: Comparison: Pregabalin vs Other Analgesics; Analysis on the mean difference between two groups with the change from baseline at Week 8; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -0.830, 95% CI 2-sided [-1.301 to -0.359]
Statistical Analysis 2: Comparison: Pregabalin vs Other Analgesics; Analysis on the mean difference between two groups with the change from baseline at Week 4; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = -0.674, 95% CI 2-sided [-1.125 to -0.223]

5. Secondary Outcome: Change From Baseline in Euro Qol 5-Dimensions (EQ-5D-5L)-QOL-Score-
Description: The EQ-5D-5L is a copyrighted, subject-completed questionnaire designed to assess health-related quality of life in terms of a single index value or utility score. The Health State Profile is designed to record the subject's level of current health for five domains comprising a health profile: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Responses from the five domains are used to calculate a single utility index value.; 1 indicates better health state (no problems); 5 indicates worst health state (eg, "confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile; from 11111 to 55555. Score is transformed and results in a total score range -0.025 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Visit2 (Week4), Final Visit (Week8 or discontinuation)
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Other Analgesics
Number analyzed (Participants) | 137 | 171
units on a scale
  Baseline (n=137,171) | 0.6647 (0.1736) | 0.7233 (0.1521)
  Change from baseline at Week 4 (n=118,158) | 0.0756 (0.0103) | 0.0427 (0.0089)
  Change from baseline at Week 8 (n=114,159) | 0.0804 (0.0113) | 0.0600 (0.0097)
Statistical Analysis 1: Comparison: Pregabalin vs Other Analgesics; Analysis on the mean difference between two groups with the change from baseline at Week 8; Test type: Superiority or Other; p = 0.175, Mixed Models Analysis; Mean Difference (Final Values) = 0.0204, 95% CI 2-sided [-0.0091 to 0.0499]
Statistical Analysis 2: Comparison: Pregabalin vs Other Analgesics; Analysis on the mean difference between two groups with the change from baseline at Week 4; Test type: Superiority or Other; p = 0.017, Mixed Models Analysis; Mean Difference (Final Values) = 0.0329, 95% CI 2-sided [0.0058 to 0.0600]

6. Secondary Outcome: Change From Baseline in Euro Qol 5-Dimensions (EQ-5D-5L)-Visual Analogue Scale -
Description: The EQ-5D-5L is a copyrighted, subject-completed questionnaire designed to assess health-related quality of life in terms of a single index value or utility score. There are two components to the EQ-5D-5L: A Health State Profile and a Visual Analogue Scale (VAS). Recent guidance suggests that the Health State Profile and VAS should be administered together.
  The Visual Analogue Scale (VAS) is designed to rate the subject's current health state on a scale from 0 to 100 where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Time Frame: Baseline, Visit2 (Week4), Final Visit (Week8 or discontinuation)
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Other Analgesics
Number analyzed (Participants) | 137 | 172
units on a scale
  Baseline (n=137,172) | 60.9 (17.63) | 63.0 (16.34)
  Change from baseline at Week 4 (n=118,159) | 2.633 (1.373) | 1.341 (1.185)
  Change from baseline at Week 8 (n=115,160) | 6.970 (1.602) | 2.272 (1.364)
Statistical Analysis 1: Comparison: Pregabalin vs Other Analgesics; Analysis on the mean difference between two groups with the change from baseline at Week 8; Test type: Superiority or Other; p = 0.026, Mixed Models Analysis; Mean Difference (Final Values) = 4.697, 95% CI 2-sided [0.552 to 8.842]
Statistical Analysis 2: Comparison: Pregabalin vs Other Analgesics; Analysis on the mean difference between two groups with the change from baseline at Week 4; Test type: Superiority or Other; p = 0.477, Mixed Models Analysis; Mean Difference (Final Values) = 1.292, 95% CI 2-sided [-2.282 to 4.866]

7. Secondary Outcome: Clinical Global Impression of Change (CGIC)
Description: The CGIC assessment includes one question (1-7 scale) inquiring about the subject's improvement considering their current disease state.; range from 1 (very much improved) to 7 (very much worse).
Time Frame: Final Visit (Week8 or discontinuation)
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Pregabalin | Other Analgesics
Number analyzed (Participants) | 125 | 163
participants
  1.Very much improved | 17 | 3
  2.Much improved | 47 | 24
  3.Minimally improved | 37 | 47
  4.No change | 24 | 79
  5.Minimally worse | 0 | 9
  6.Much worse | 0 | 1
  7.Very much worse | 0 | 0
Statistical Analysis 1: Comparison: Pregabalin vs Other Analgesics; Test type: Superiority or Other; p < 0.001, Modified Chi-squared

8. Secondary Outcome: Patient Global Improvement of Change (PGIC)
Description: The PGIC is a subject-rated instrument that measures change in the subject's overall status on a 7-point scale. Scores range from 1 (very much improved) to 7 (very much worse).
Time Frame: Final Visit (Week8 or discontinuation)
Population: Full Analysis Set
Measure: Number; unit: participants
Groups:
- Pregabalin: 1.Patients will be treated for 8 weeks with pregabalin in primary care:no intervention
- Other Analgesics: 2.Patients will be treated for 8 weeks with other analgesics in usual care:no intervention
Arm/Group | Pregabalin | Other Analgesics
Number analyzed (Participants) | 117 | 161
participants
  1.Very much improved | 8 | 5
  2.Much improved | 34 | 22
  3.Minimally improved | 45 | 44
  4.No change | 27 | 71
  5.Minimally worse | 3 | 17
  6.Much worse | 0 | 1
  7.Very much worse | 0 | 1
Statistical Analysis 1: Comparison: Pregabalin vs Other Analgesics; Test type: Superiority or Other; p < 0.001, Modified Chi-squared

9. Secondary Outcome: Work Productivity and Activity Impairment Scale (WPAI:LBP)
Description: The WPAI: LBP is a self-administered questionnaire that measures the effect of general health and symptom severity on work productivity and regular activities. Subscale scores include Percent work time missed due to pain (PWP), Percent overall work impairment (PWI), Percent work productivity impairment due to pain (PWPI), Percent overall activity impairment (PAI). Each subscale score is expressed as an impairment percentage (0-100) where higher numbers indicate greater impairment and less productivity. Here, "n" signifies "Number of participants" for Baseline.
  In this study, the WPAI: LBP will measure the effect of the patient's Chronic Low Back Pain (CLBP) with accompanying lower limb pain (neuropathic component) on work productivity and regular activities.
Time Frame: Final Visit (Week8 or discontinuation)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of time missed
Groups:
- Other Analgesics: Patients will be treated for 8 weeks with other analgesics in usual care : no intervention
Arm/Group | Pregabalin | Other Analgesics
Number analyzed (Participants) | 137 | 172
percentage of time missed
  1.PWP (n=43, 56) | 0.13 (0.863) | 1.61 (7.574)
  2.PWI (n=43, 55) | 28.84 (23.726) | 27.09 (24.771)
  3.PWPI (n=43, 55) | 28.88 (23.797) | 27.84 (25.814)
  4.PAI (n=42, 56) | 31.19 (26.152) | 29.64 (23.039)

10. Other Pre Specified Outcome: Number of Patients With Adverse Events
Time Frame: Visit2(week4),Final Visit(Week8 or discontinuation)
Population: Safety Analysis Set; All subjects who received at least one dose of pregabalin. The primary objectives of this study did not include comparison of safety with usual care, consistent with the non-interventional nature of the study. Therefore, adverse events were not collected from the participants in usual care.
Measure: Number; unit: participants of related AEs
Groups:
- Pregabalin: Patients will be treated for 8 weeks with pregabalin in primary care : No intervention
Arm/Group | Pregabalin
Number analyzed (Participants) | 157
participants of related AEs | 56

ADVERSE EVENTS:
Time Frame: Baseline to Week 4, Week 8
Description: Safety Analysis Set; All subjects who received at least one dose of pregabalin. The primary objectives of this study did not include comparison of safety with usual care, consistent with the non-interventional nature of the study. Therefore, adverse events were not collected from the participants in usual care.
Groups:
- Pregabalin: Patients will be treated for 8 weeks with pregabalin in primary care No intervention: The study is observational
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 0/157
Other Adverse Events (participants affected / at risk) | 40/157
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=157)
Nausea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 17 (17)
Headache (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No